CLINICAL TRIAL: NCT03595735
Title: The Zenflow Spring System Safety, Performance and Effectiveness Study (ZEST2)
Brief Title: The Zenflow Spring System Safety, Performance and Effectiveness Study
Acronym: ZEST2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zenflow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0043
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, single-arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Receives treatment with the Zenflow Spring System
  Interventions: Device: Zenflow Spring System

INTERVENTIONS:
Device: Zenflow Spring System — The Zenflow Spring System consists of the Spring Delivery System with Implant, Spring Scope, Camera Control Unit (CCU), Measurement Tool, and Spring Retrieval Tool.
  Other Names: Spring Implant

SUMMARY:
This is a clinical evaluation to assess the safety and performance of the Zenflow Spring System when used as intended to relieve symptoms of obstructive Benign Prostatic Hyperplasia (BPH).

DETAILED DESCRIPTION:
A multi-center, prospective, single arm safety, performance, and effectiveness trial. The study will be conducted in two stages. Upon the successful completion of stage 1, the study will be expanded and continue to stage 2.

Stage 1 will enroll subjects in the Intent to Treat (ITT) cohort. The purpose of stage 1 is to assess acute safety and performance of the Zenflow System at the time of the procedure, through discharge, 2 weeks and 1 month, in up to 10 subjects enrolled at up to 7 investigational sites, to determine continuation to stage 2.

Upon successful completion of stage 1, the study will be expanded to stage 2 with sites added and continued enrollment in the ITT cohort. All subjects, including those enrolled in the stage 1 evaluation, will continue to be followed at all the designated follow-up time points for the full duration of the study (60 months).

Whether or not the study continues to Stage 2, all enrolled subjects will be followed for the entire duration of the study (60 months), or until exited.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to meet the following inclusion criteria in order to be considered eligible for participation in this trial:

1. ≥ 45 years of age
2. Baseline IPSS score > 13, and a baseline Quality of Life (QoL) question score > 3
3. Prostate volume 25 - 80 cc by Trans Rectal Ultrasound (TRUS), measured within past 90 days and prostatic urethral length between 2.5-4.5 cm.
4. Failed or intolerant to medication regimen for the treatment of LUTS.

Exclusion Criteria:

Subjects will be excluded from participating in this trial if they meet any of the following criteria:

1. Obstructive intravesical median prostatic lobe or high bladder neck
2. Urethral stricture, meatal stenosis, or bladder neck obstruction - either current, or recurrent requiring 2 or more dilatations
3. Baseline PSA > 10 ng/mL or confirmed or suspected prostate cancer
4. Elevated risk of prostate cancer
5. Post-void residual volume (PVR) > 250 ml
6. Peak urinary flow rate > 12 ml/second, with ≥ 125 ml voided volume at baseline
7. History of chronic urinary retention
8. History of neurogenic bladder
9. Compromised renal function (e.g., serum creatinine > 1.8 mg/dl) due to bladder obstruction
10. Concomitant Urinary Tract Infection (UTI) (subject can be enrolled following successful treatment of UTI and a clean urine test)
11. Concomitant bladder stones
12. Confirmed or suspected bladder cancer
13. Previous pelvic irradiation or radical pelvic surgery
14. Previous prostate surgery, stent implantations, laser prostatectomy, hyperthermia or another invasive treatment to the prostate
15. Chronic prostatitis, or recurring prostatitis within the past 12 months
16. Serious concurrent medical conditions such as uncontrolled diabetes
17. Known allergy to nickel
18. Life expectancy less than 24 months
19. Use of concomitant medications (e.g., anticholinergics, antispasmodics or antidepressants) affecting bladder function
20. Patients taking coumadin 3 days or less prior to procedure and have INR value > 1.5 on day of procedure. ASA and clopidogrel must be ceased 7 days prior to the procedure
21. 5 alpha reductase inhibitors within 6 months of pre-treatment evaluation unless evidence of same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued for entrance into or throughout the study)
22. alpha blockers within 2 weeks of pre-treatment evaluation unless evidence of same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued for entrance into or throughout the study)
23. Future fertility concerns
24. Any severe illness that might prevent study completion or would confound study results

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Successful placement of the Zenflow Spring Implant | Day of discharge up to 7 days following device placement
  Successful deployment and procedural success for the Zenflow System to implant the Spring device in the operating room or an out-patient clinical setting.
Need for urinary catheterization | 7 days after the procedure
  Rate of extended post-operative urinary catheterization

SECONDARY OUTCOMES:
Incidence of procedure or device related serious adverse events | Day of discharge up to 7 days following device placement
  Assessment of any device or procedure related Serious Adverse Events (SAE)
Assessment of Pain | Baseline, 2 weeks, 1 month and 3 months
  Patient describes pain on a Visual Analog Scale (VAS). The scale is a line labeled 1 at the far left indicating minimal pain and 10 on the right, which is maximum pain.
Assessment of Adverse Events | Up to 2 years
  Rate of adverse events related to the procedure or device.
Assessment of Sexual Health: Change in sexual health measured by change in the Sexual Health Inventory for Men (SHIM) questionnaire score | Baseline, 3, 6, 12, & 24 months
  The patient selects the most appropriate response to 5 questions about his sexual health. Each response has an assigned value between 1 and 5. The numeric values are tallied for a total score.
Assessment of Sexual Health: Change in sexual health measured by change in ability to ejaculate using the Male Sexual Health Questionnaire - Ejaculatory domain (MSHQ-EjD) | Baseline, 3, 6, 12, & 24 months
  The patient selects the most appropriate response to 4 questions about his sexual health specific to ejaculation. Each response has an assigned value between 0 and 5.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) by patient response to the International Prostate Symptom Score and Quality of Life Questionnaire (IPSS+QoL). | Baseline, 2 weeks, 1, 6, 12, 24 months
  The patient is asked to respond to 7 questions related to his urinary health using a rating scale of 0 to 5 where is zero is excellent and 5 is the worst possible. The responses to the 7 questions are tallied for a total score. In addition the patient is asked 1 question related to his Quality of Life. The possible responses range from 0 to 6 where 0 is the best and 6 is the worst.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) | Baseline, 2 weeks, 1, 3, 6, 12, 24 months
  Improvement in flow of urine
Repeat interventions to treat Benign Prostatic Hyperplasia (BPH) | Up to 2 years
  Incidence of repeat invasive treatment for Lower Urinary Tract Symptoms (LUTS) or increase in dosage or initiation of new medication to treat symptoms of BPH.
Increase or change in medications to treat Benign Prostatic Hyperplasia (BPH) | Up to 2 years
  Incidence of increase in dosage, or initiation of new medication to treat symptoms of BPH.

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Galan, MD, Principal Investigator — Centro de Urología Avanzada del Noreste (CUAN)
Locations (3):
- Mexico (3):
  - Hospital Regional de Alta Especialidad de Ixtapaluca, Zoquiapan, Ciudad de Ixtapaluca
  - Hospital Universitario "Dr. José Eleuterio González", Monterrey, Nuevo León
  - Centro de Urología Avanzada del Noreste (CUAN), Monterrey, Nuevo León